CLINICAL TRIAL: NCT00458458
Title: Treatment of Endometriosis With Norethindrone Acetate ( NA) VS. Gonadotropin- Releasing Hormone (GnRH) Agonist (Lupron Depot 11.25 mg)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: State University of New York - Downstate Medical Center (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ozgul Muneyyirci-Delale, Director of Division of Reproductive Endocrinology and Infertility, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HD043281 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-10 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Endometriosis; Dysmenorrhea; Dyspareunia
Keywords: Endometriosis; Dysmenorrhea; Pelvic Pain; Period Pain; Menstrual Cramps; Dyspareunia; Norethindrone Acetate; Lupron Depot; Bone Density; Lipid Profile
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Dyspareunia; Pelvic Pain | interventions — Norethindrone Acetate; Gonadotropin-Releasing Hormone; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NA alone (Active Comparator): Norethindrone Acetate (NA) 5mg taken 1-3 tabs orally every night for duration of treatment
  Interventions: Drug: Norethindrone Acetate (NA)
- LD then NA (Active Comparator): Lupron Depot(LD) given intramuscularly every 12 weeks for total of 24 weeks then switched to Norethindrone Acetate (NA) taken 1-3 tablets orally every night for remainder of treatment
  Interventions: Drug: GnRH Agonist (Lupron Depot)

INTERVENTIONS:
Drug: Norethindrone Acetate (NA) — 52 weeks of treatment with Norethindrone Acetate
  Arms: NA alone
Drug: GnRH Agonist (Lupron Depot) — 24 weeks of treatment with Lupron Depot then 28 weeks of treatment with Norethindrone Acetate
  Arms: LD then NA

SUMMARY:
(A) Major 1) to compare the effectiveness of norethindrone acetate (NA) with GnRH agonist (Lupron-Depot-3) in relieving symptoms of endometriosis, 2) to compare bone density in the two treated groups in order to demonstrate that NA does not affect bone density; (B) Minor: 1) To compare the lipid profiles of patients in the two groups to confirm the hypothesis that the effects of NA and GnRH agonists on lipid profiles are similar, 2) To determine whether quality of life, assessed by questionnaire, is better in patients assigned to NA than in patients assigned to GnRH, 3) To determine whether NA has fewer adverse effects than GnRH agonist.

DETAILED DESCRIPTION:
Objectives: (A) Major 1) to compare the effectiveness of norethindrone acetate (NA) with GnRH agonist (Lupron-Depot-3) in relieving symptoms of endometriosis, 2) to compare bone density in the two treated groups in order to demonstrate that NA does not affect bone density; (B) Minor: 1) To compare the lipid profiles of patients in the two groups to confirm the hypothesis that the effects of NA and GnRH agonists on lipid profiles are similar, 2) To determine whether quality of life, assessed by questionnaire, is better in patients assigned to NA than in patients assigned to GnRH, 3) To determine whether NA has fewer adverse effects than GnRH agonist.

After signing an IRB approved consent from 112 women with symptomatic endometriosis, diagnosed surgically, will be treated with NA or Lupron-Depot-3 for 24 weeks. After 24 weeks both groups will be treated only with NA until 52 weeks. After that, both groups will be followed for an additional 52 weeks to assess any return of clinical symptoms and to determine whether laboratory tests of drug related changes return to pretreatment levels.

Treatment regimens are as follows: For the first 24 weeks, women in the NA group will be treated with 5 mg NA daily and a placebo injection every 12 weeks. In case of bleeding, the NA dose will be increased (max 15 mg) until bleeding stops, and then decreased by 2.5 mg every 4 weeks to a final dose of 7.5 mg which will be maintained for the remainder of the 24 weeks. For the first 24 weeks, women in the GnRH groups will receive Lupron-Depot-3 injections every 12 weeks plus placebo pills daily - bleeding will be treated with an increase in placebo pills to simulate treatment in the NA group. After 24 weeks, all women will be on identical regimens of 5 mg NA pills daily and no injections.

On the first treatment day, subjects will have the following tests/assessments: bone density with DEXA, scoring of endometriosis symptoms, quality of life questionnaire, general physical examination, lipid profile, estradiol (E2), N-telopeptide, and pregnancy test. All tests, except bone density and lipid profile, will be repeated at 12, 24, and 52 weeks of treatment. Bone density will be performed at 24 and 52 weeks and lipid profile will be performed at 12 and 52 weeks of treatment. In the follow-up period, physical examination, quality of life questionnaires, scoring of symptoms will be done at 3, 6, 9 and 12 months. Lipid profile, N-telopeptide and E2 will be performed at 3 and 12 months and bone density at 12 month follow-up.

The objectives stated above will be compared between the two groups at 12, 24, and 52 weeks of treatment and at 6-month intervals during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The subject has voluntarily signed the Informed Consent form after having the contents fully explained, after all questions are answered and prior to undergoing any study-related procedures.
* The subject is a pre-menopausal female at least 18 years of age at the time of screening having regular periods (21-42 days intervals) with no menopausal symptoms.
* The subject has a diagnosis of endometriosis made via laparoscopy or laparotomy (operative report will be obtained) and still symptomatic and at least 3 months after surgery have a grade 2 and above according to Biberoglu's pain grade at screening visit (4 weeks prior initiation of treatment) or 4 out of 10 on a visual pain scale (visual analogue)
* Subject in good health, except for endometriosis, or has mild medical conditions that are stable and controlled. The subject has no clinically relevant hepatic, renal, cardiovascular, respiratory, endocrine, metabolic, psychiatric, neurologic (epilepsy), hematolytic (coagulopathy) and/or immunologic disease (on steroids) or disorder.
* A subject who has received any of the hormone therapies (GnRH agonist or danazol or progestin) must meet the minimum washout requirement to be eligible. (GnRH within the last 6 months and with steroids within the last month.) After hormonal therapy has stopped, the subject must have returned to normal for at least two menstrual cycles before baseline time.
* Serum pregnancy and urine qualitative pregnancy tests performed at screening and on baseline must be negative.
* Unless surgical sterile by bilateral tubal ligation or vasectomy of partner, the subject agrees to use a double-barrier method of contraception during the screening period, throughout the 24-week treatment period, such as: condom plus spermicide, diaphragm plus spermicide, sponge plus spermicide, abstinence is an acceptable form of birth control.
* Less than grade III overweight or BMI <40 kg/M2

Exclusion Criteria:

* Less than 3 months postpartum and post-lactation at the time of dosing.
* Abnormal laboratory findings considered clinically significant if more than twice the normal range. Abnormal tests will be repeated, and if still high as stated before, subject will be excluded.
* A previous history of significant adverse reactions to hormone, progestin or progesterone and GnRH agonist therapies.
* Abnormal Pap smear in the last 6 months. Subjects with ASCUS (atypical squamous cells of undetermined significance) and are negative for high-risk human papilloma virus (HPV) will be eligible. Subjects that have atypical endocervical cells, and atypical glandular cells are not eligible for this study.
* Subject has a bone density T score less or equal to 2.5, history of nontraumatic fracture, history of spinal surgery, history of fusion of lumbar region, history of severe scoliosis greater than 20 degrees.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2004-08; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of norethindrone acetate (NA) with GnRH agonist (Lupron-Depot-3) in relieving symptoms of endometriosis | First 24 weeks of treatment
To compare effect of norethindrone acetate (NA) with GnRH agonist (Lupron-Depot-3)on bone density | 52 weeks of treatment
  Bone density with be compared in the two treated groups in order to demonstrate that NA does not affect bone density.

SECONDARY OUTCOMES:
To compare the effect of norethindrone acetate (NA) with GnRH agonist (Lupron-Depot-3)on lipid profiles | Treatment and follow-up
  Lipid profiles of patients in the two groups will be collected to confirm the hypothesis that the effects of NA and GnRH agonists on lipid profiles are similar.
To determine the effect treatment has on quality of life | Treatment and follow-up
  Quality of life will be assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ozgul Muneyyirci-Delale, M.D., Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States